CLINICAL TRIAL: NCT05628649
Title: Teaching Kitchen Multisite Trial (TK-MT)
Brief Title: Teaching Kitchen Multisite Trial
Acronym: TKMT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: Teaching Kitchen Collaborative, Inc. (Unknown); University of California, Los Angeles (Other); University of California, Irvine (Other); The University of Texas Health Science Center, Houston (Other); Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Dr. Jennifer Susan Massa, Study Implementation Leader, Harvard School of Public Health (HSPH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB22-0506
Record Dates: First submitted 2022-07-27; First posted 2022-11-29 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Experimental): Participants in the intervention group will gather together in a 2-hour group setting once a week for the first 16 week intensive, then change to a once a month 2-hour gathering for the remaining 8 months of boosters of the intervention. Follow-up will occur 6 months after the final intervention class to assess long-term changes. The total time span of the study will be 18 months.
  Interventions: Behavioral: Teaching Kitchen Collaborative Curriculum
- Control (No Intervention): The control group follows clinical care in the usual standard (i.e. continuing to receive usual care from one's primary care physician)

INTERVENTIONS:
Behavioral: Teaching Kitchen Collaborative Curriculum — Participants in the intervention arm will first attend 16 weeks of intensive 2-hour classes covering hands-on cooking skills, dietary recommendations (as described within the Harvard Healthy Eating Plate), mindfulness and stress reduction skills, activity and movement techniques, and tools for behavior change. Next, they will attend monthly booster classes for 8 months, with a final assessment for the sustainability of outcomes at 18 months. Sessions will be taught by a combination of a chef educator, dietitian, health coach, or medical doctor.
  The study will consist of 2 cohorts of individuals from 4 teaching kitchen program institutions. Each institution will run one-two cycles of the program with each cycle including both a treatment and control group. Each individual cohort will consist of a maximum of 80 individuals; with 40 block-randomized to the intervention and 40 in the control group receiving normal standard of care (followed by their PCP).
  Arms: Intervention

SUMMARY:
This TK-MT is an interactive year-long program that teaches culinary skills, nutrition education, mindfulness, and stress reduction, promotes movement, and optimizes behavior change through health coaching strategies. The purpose of this study is to test whether a referral-based teaching kitchen intervention offered for 12 months in adjunct to primary care obesity management is feasible, acceptable, and effective on improving health behaviors and obesity prevention. Specifically, the primary goal of the study is to provide evidence of improved behavior change (ex: increases in cooking at home, fruit and vegetable intake, exercise, sleep, mindful activities), improved lab values (ex: fasting blood glucose, cholesterol, triglycerides, etc.), and resulting change in body weight and waist circumference measures. The hypothesis is that by participating in this novel TK-MT intervention - learning to cook healthy, delicious, inexpensive meals at home; understanding principles of good nutrition (based on the Harvard Healthy Eating Plate); incorporating exercise more effectively into daily living; reducing stress and increasing mindfulness and sleep; and, having access to principles of health coaching - in order to leverage personal motivations - can provide a platform to transform individuals and consequently their health, not only for the duration of this study (16 weeks intensive, 8 months boosters for a total of 12 months) but for their entire lives.

ELIGIBILITY:
Inclusion Criteria:

* Capacity for consent
* Adults living independently
* English literate
* Aged 25-70 (to capture adults living independently)
* Diagnosis of class I or II obesity (BMI 30-39.9 kg/m2)
* Abnormality in one of the following metabolic markers (fasting plasma concentrations of glucose, insulin, ALT/AST and lipids including cholesterol, triglycerides, LDL, or HDL)
* Available and willing to commit to the 18 month study including: 16 consecutive weekly classes; 8 once a month classes; along with assessments at 0, 4, 12, and 18 months.

  * Participants must be able to commit to both in person and virtually participation
* Access to two devices, one device with a camera (smartphone, tablet, computer)
* Reliable internet connect in their home

  * Capable of operating device independently
* Minimal operational cooking appliances; specifically cooktop and oven at home.

Biometric and Anthropometric Markers:

* Fasting glucose - minimum: 100 mg/dL; maximum: 125 mg/dL
* Hemoglobin A1C - minimum: 5.7% maximum: 6.4%
* Triglycerides - minimum: 150 mg/dL; maximum: 500 mg/dL
* LDL - minimum: 130 mg/dL; maximum: 190 mg/dL
* HDL - minimum: men < 40 mg/dL; women < 50 mg/dL
* LDL/HDL ratio - minimum: men > 3.0; women > 2.5
* Blood Pressure - minimum: systolic 130 mmHg and diastolic <80 mmHg; maximum: uncontrolled HTN per PCP
* Waist Circumference - minimum: men > 94 cm; women > 80 cm
* ALT - minimum: men > 55 unit/L; women > 30 unit/L; maximum: 4x limit

Exclusion Criteria:

* Anaphylactic reaction to food allergens
* Relocating out of area in the next 18 months
* Taking obesity or diabetes medication (with the exception of metformin) as assessed by the study medical director
* Current or past diagnosis of Type 1 or 2 diabetes (excluding past gestational diabetes)
* History of severe obesity (BMI>=40kg/m2)
* History of bariatric surgery
* Current or planned (during study period) participation in a formal longitudinal culinary or weight management program at the time of recruitment (ie-any smart phone apps, a virtual classes, or in person classes or coaching)
* Psychiatric hospitalization in the past 12 months
* History of significant mental health diagnoses or recent life-threatening illnesses (including unstable cardiovascular disease)
* Alcohol or substance abuse within the past 12 months
* Diet / exercise contraindications to program participation
* Other medical, psychiatric, or behavioral limitations that in the judgment of the principal investigator or study site PI's may interfere with study participation or the ability to follow the intervention protocols determined by each site's PI
* Prisoners, pregnant women, and women planning to become pregnant over the next 18 months
* Unable or unwilling to give informed consent or communicate per protocol with local study staff
* Unwilling or unable to participate in all study-related activities

Ages: 25 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Program feasibility based on number referred | first 3 months
  Number of completed referrals received
Program feasibility based on referral rate | first 3 months
  Calculated using the following formula: (# enrolled / # referred)
Program feasibility based on number enrolled | first 3 months
  number of participants enrolled in the study
Program feasibility based on enrollment rate | first 3 months
  Calculated using the following formula: [# enrolled / (# referred & eligible)].
Program feasibility based on eligible but not enrolled | first 3 months
  Number of people eligible but not enrolled and reason
Change in program attendance | at each of the 16 weekly intensive sessions followed by 8 monthly booster sessions
  The number of classes participants attend is counted as program attendance. This outcome will be measuring program feasibility based on program attendance
Program feasibility based on program completion | at 12 months
  Number completing program (defined as >80% of sessions)
Change in completion rate over time | at each of the 16 weekly intensive sessions followed by 8 monthly booster sessions
  Completion rate is calculated using the following formula: (# completing all classes / # enrolled). This outcome will be measuring program feasibility based on completion rate.
Program feasibility based on acceptable completion rate | at 12 months
  Calculated using the following formula: (>75% sessions / # enrolled)
Change in assessment completion rate | at each of the 16 weekly sessions, 4 months follow-up, each of the 8 monthly sessions, 12 months follow up, and 18 months follow-up
  Assessment completion rate is calculated using the following formula: (# completing all assessments / # enrolled). This outcome will be measuring program feasibility based on assessment completion rate.
Program Feasibility based on the number of screen failures | first 3 months
  Number of people referred but not eligible and reason
Program feasibility based on number of withdrawals (dropouts) | at 18 months (per each cohort)
  Number of enrolled participants officially withdrawing from the study and reason for withdrawal
Program feasibility based on number lost to follow up (attrition) | at 6 months (per each cohort)
  Number who failed to attend sessions and could not be contacted for follow-up
Program acceptability based on qualitative components from participant interviews. | after the final class session at 12 months or during month 13
  This outcome measures program acceptability based on qualitative components from participant interviews.
  Thematic analysis will be conducted by the central Harvard team through transcriptions via qualitative analysis software using open and then focused coding. We may use iScribed.com (or approved service) and Dedoose or similar programs for transcription and analysis of the interviews.
Program acceptability based on staff interviews. | after the final class session at 12 months or during month 13
  This outcome measures program acceptability based on qualitative components from staff interviews.
  Thematic analysis will be conducted by the central Harvard team through transcriptions via qualitative analysis software using open and then focused coding. We may use iScribed.com (or approved service) and Dedoose or similar programs for transcription and analysis of the interviews.
Change in program acceptability based on open-ended survey items for participants. | baseline, 4 months, 12 months, and 18 months
  This outcome measures the change in program acceptability based on qualitative components from open-ended survey items.
  Thematic analysis will be conducted by the central Harvard team through transcriptions via qualitative analysis software using open and then focused coding. We may use iScribed.com (or approved service) and Dedoose or similar programs for transcription and analysis of the interviews.
Change in program acceptability based on post-class surveys. | after each of the 16 weekly intensive sessions followed by the 8 monthly booster sessions.
  This outcome is measuring the change in program acceptability based on quantitative components from post-class surveys. Specifically, change in participant satisfaction and experience using a [1-5] Likert scale (1 being a less favorable response, and 5 is a more favorable response) will be collected.
  Descriptive statistics (means, medians, proportions, 95% confidence intervals [CI]) will be computed and data will be analyzed to assess for change. A paired t-test will evaluate pre/post changes in continuous measures.
Change in program acceptability based on other quantitative survey items addressing participant satisfaction. | at each of the 16 weekly intensive sessions, 4 months follow-up, each of the 8 monthly booster sessions,12 months follow-up, and 18 months follow-up
  This outcome is measuring the change in program acceptability based on quantitative components from other quantitative surveys addressing participant satisfaction.
  Descriptive statistics (means, medians, proportions, 95% confidence intervals [CI]) will be computed and data will be analyzed to assess for change. A paired t-test will evaluate pre/post changes in continuous measures.
Change in the fidelity of program implementation based on participant interview. | after the final class session at 12 months or during month 13
  Semi-structured interviews with participants will evaluate barriers and facilitators to meeting participant needs, perceived need for innovation, and participant feedback.
  Qualitative Measures: Thematic analysis will be conducted by two researchers who will independently read transcripts and conduct open and then focused coding. Open-ended questionnaire items will also assess the TK participant assessment tool and be included for qualitative data. iScribed.com and Dedoose or similar programs might be used for transcription and analysis of the interviews.
Change in the fidelity of program implementation based on open-ended survey items for participants. | baseline, 4 months, 12 months, and 18 months
  This outcome measures the change in the fidelity of program implementation based on barriers and facilitators reported by participants via open-ended survey items.
  Qualitative Measures: Thematic analysis will be conducted by two researchers who will independently read transcripts and conduct open and then focused coding. Open-ended questionnaire items will also assess the TK participant assessment tool and be included for qualitative data.
Change in the opinion on the TK assessment tool. | baseline and 4 months
  This outcome measures the change in the fidelity of program implementation based on a quantitative participant questionnaire used to collect feedback on the TK assessment tool.
  Participants will complete a questionnaire to elicit feedback on the TK assessment tool. This quantitative questionnaire will collect binary and likert-scale based responses. The responses in the questionnaire in totality will be used to calculate the change in opinion.
Socioeconomic determinants of health | baseline
  Socioeconomic determinants of health information from participant demographics

SECONDARY OUTCOMES:
Change in TK participant assessment results | baseline, 4, 12, and 18 months
  The TK participant assessment is an investigator-created, non-validated Health Habits Survey that assesses nutrition, exercise, cooking habits, sleep behaviors, basic medical information, readiness to change, mindfulness, and telehealth experience. Individual survey questions have variable response categories. For example, commitment to change is assessed using a 1 to 10 scale with 1 being a less favorable response, and 10 is a more favorable response.
Change in nutrition or dietary consumption and patterns as measured by Modified PDQS-30 days assessment | baseline, 4, 12, and 18 months
  measured by participants' self-reported eating habits on fruits, vegetables, and other diet habits. Scores associated with the healthier dietary pattern are higher and lower for unhealthy patterns.
Change in movement and exercise as measured by exercise vital sign (EVS) | baseline 4, 12, and 18 months
  EVS is calculated by multiplying responses to "On average, how many days per week do you engage in moderate to strenuous exercise (like a brisk walk)?" and "On average, how many minutes per day do you engage in exercise at this level?" in order to display minutes per day of moderate or strenuous exercise.
Change in the quality and amount of sleep as measured by APA DSM5 | baseline 4, 12, and 18 months
  The Patient-Reported Outcomes Measurement Information System (PROMIS) Sleep Disturbance instruments assess self-reported perceptions of sleep quality, sleep depth, and restoration associated with sleep. This includes perceived difficulties and concerns with getting to sleep or staying asleep, as well as perceptions of the adequacy of and satisfaction with sleep.
Change in mindfulness, in general, and as applied to eating and cooking as measured by FMI Mindfulness Questionnaire | baseline, 4, 12 and 18 months
  The Freiburg Mindfulness Inventory (FMI) is an instrument that assesses mindfulness.
Change in readiness-to-change as measured by the University Rhode Island Change Assessment Scale (URICA): Short Form for Physical Health Behavior State | baseline, 4, 12 and 18 months
  Self-reported survey of respondents' feelings about changing their weight problem. Total score is also called the Readiness Score, ranging from -2 to +14 (worse to better), calculated by subtracting the mean from the precontemplation responses from the summation of the means of responses to contemplation, action, and the struggling to maintain items.
Cooking frequency and competency using existing assessment tools as well as additional single survey items to enhance assessment | baseline, 4, 12 and 18 months
  Self Efficacy for Eating/Cooking Fruit and Vegetables assessment by Condrasky: Cooking attitudes as measured by self-reported attitudes about cooking and the use of the provided fresh fruits and vegetables to provide food to themselves and or their families.
Change in quality of life, quality of work-life balance as measured by RAND 20-Item Short Form Health Survey | baseline, 4, 12 and 18 months
  Quality of life will be assessed using the 20-item Short Form Survey Instrument (SF-20). It was developed by the RAND corporation. The SF-20 is a well accepted and valid survey used to assess overall health measuring 8 different dimensions including physical and social functionality and limitations, mental health, vitality, pain, general health perception, and health change
Change in cooking frequency as measured by Gallup Poll cooking frequency questionnaire | baseline, 4, 12 and 18 months
  The cooking frequency questionnaire measures the frequency of eating and cooking lunch or dinner at home in the past week.
Overall rating and impressions of the class session as measured by class feedback survey. | at the conclusion of each of the 16 weekly intensive sessions and 8 monthly booster sessions
  Class feedback survey will assess the overall rating and impressions of the class session.
Change in Fasting glucose | baseline, 4, 12 and 18 months
  Fasting glucose (mg/dL)
Change in Fasting Insulin | baseline, 4, 12 and 18 months
  Fasting insulin (mg/dL)
Change in Fasting Lipid Profile | baseline, 4, 12 and 18 months
  total cholesterol (mg/dL), triglycerides (mg/dL), HDL (mg/dL) and LDL (mg/dL)
Change in Hemoglobin A1c | baseline, 4, 12 and 18 months
  Hemoglobin A1c mmol/mol
Change in ALT | baseline, 4, 12 and 18 months
  Hemoglobin ALT (mg/dL)
Change in Systolic Blood Pressure | baseline, 4, 12 and 18 months
  Blood pressure (mmHg)
Change in Diastolic Blood Pressure | baseline, 4, 12 and 18 months
  Blood pressure (mmHg)
Change in body weight | at baseline, each of the 16 weekly intensive sessions, 4 months follow-up, each of the 8 monthly booster sessions, 12 months follow-up, and 18 months follow-up
  Body weight will be measured (kg)
Change in Body Mass Index | baseline, 4, 12 and 18 months
  Height (cm) and Weight (kg) will be used to calculate body mass index (kg/m^2)
Change in Waist Circumference | baseline, 4, 12 and 18 months
  Waist circumference will be measured (cm)

CONTACTS AND LOCATIONS:
Overall Officials: Kate Janisch, MPH, RDN, Study Director — HSPH
Locations (5):
- United States (5):
  - University of California Irvine, Irvine, California
  - University of California Los Angelos, Los Angeles, California
  - Harvard Coordinating Site, Boston, Massachusetts
  - Dartmouth Health, Lebanon, New Hampshire
  - UTHealth Houston, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] CDC. Chronic Diseases in America. Centers for Disease Control and Prevention. Published May 6, 2022. Accessed June 5, 2022. https://www.cdc.gov/chronicdisease/resources/infographic/chronic-diseases.htm
- [Background] Schwingshackl L, Hoffmann G, Lampousi AM, Knuppel S, Iqbal K, Schwedhelm C, Bechthold A, Schlesinger S, Boeing H. Food groups and risk of type 2 diabetes mellitus: a systematic review and meta-analysis of prospective studies. Eur J Epidemiol. 2017 May;32(5):363-375. doi: 10.1007/s10654-017-0246-y. Epub 2017 Apr 10. PMID 28397016
- [Background] Chanson-Rolle A, Meynier A, Aubin F, Lappi J, Poutanen K, Vinoy S, Braesco V. Systematic Review and Meta-Analysis of Human Studies to Support a Quantitative Recommendation for Whole Grain Intake in Relation to Type 2 Diabetes. PLoS One. 2015 Jun 22;10(6):e0131377. doi: 10.1371/journal.pone.0131377. eCollection 2015. PMID 26098118
- [Background] Eisenberg DM, Righter AC, Matthews B, Zhang W, Willett WC, Massa J. Feasibility Pilot Study of a Teaching Kitchen and Self-Care Curriculum in a Workplace Setting. Am J Lifestyle Med. 2017 May 23;13(3):319-330. doi: 10.1177/1559827617709757. eCollection 2019 May-Jun. PMID 31105496
- [Background] Dasgupta K, Hajna S, Joseph L, Da Costa D, Christopoulos S, Gougeon R. Effects of meal preparation training on body weight, glycemia, and blood pressure: results of a phase 2 trial in type 2 diabetes. Int J Behav Nutr Phys Act. 2012 Oct 17;9:125. doi: 10.1186/1479-5868-9-125. PMID 23075398
- [Background] Ricanati EH, Golubic M, Yang D, Saager L, Mascha EJ, Roizen MF. Mitigating preventable chronic disease: Progress report of the Cleveland Clinic's Lifestyle 180 program. Nutr Metab (Lond). 2011 Nov 23;8:83. doi: 10.1186/1743-7075-8-83. PMID 22112436
- [Background] Shepherd E, Gomersall JC, Tieu J, Han S, Crowther CA, Middleton P. Combined diet and exercise interventions for preventing gestational diabetes mellitus. Cochrane Database Syst Rev. 2017 Nov 13;11(11):CD010443. doi: 10.1002/14651858.CD010443.pub3. PMID 29129039
- [Background] World Health Organization. Notes for the media: New physical activity guidance can help reduce risk of breast, colon cancers; 2011. Accessed January 28, 2012.
- [Background] Katterman SN, Kleinman BM, Hood MM, Nackers LM, Corsica JA. Mindfulness meditation as an intervention for binge eating, emotional eating, and weight loss: a systematic review. Eat Behav. 2014 Apr;15(2):197-204. doi: 10.1016/j.eatbeh.2014.01.005. Epub 2014 Feb 1. PMID 24854804
- [Background] Ammentorp J, Uhrenfeldt L, Angel F, Ehrensvard M, Carlsen EB, Kofoed PE. Can life coaching improve health outcomes?--A systematic review of intervention studies. BMC Health Serv Res. 2013 Oct 22;13:428. doi: 10.1186/1472-6963-13-428. PMID 24148189
- [Background] Kronsteiner-Gicevic S, Mou Y, Bromage S, Fung TT, Willett W. Development of a Diet Quality Screener for Global Use: Evaluation in a Sample of US Women. J Acad Nutr Diet. 2021 May;121(5):854-871.e6. doi: 10.1016/j.jand.2020.12.024. Epub 2021 Feb 15. PMID 33602635
- [Background] Coleman KJ, Ngor E, Reynolds K, Quinn VP, Koebnick C, Young DR, Sternfeld B, Sallis RE. Initial validation of an exercise "vital sign" in electronic medical records. Med Sci Sports Exerc. 2012 Nov;44(11):2071-6. doi: 10.1249/MSS.0b013e3182630ec1. PMID 22688832
- [Background] Yu L, Buysse DJ, Germain A, Moul DE, Stover A, Dodds NE, Johnston KL, Pilkonis PA. Development of short forms from the PROMIS sleep disturbance and Sleep-Related Impairment item banks. Behav Sleep Med. 2011 Dec 28;10(1):6-24. doi: 10.1080/15402002.2012.636266. PMID 22250775
- [Background] Walach H, Buchheld N, Buttenmüller V, Kleinknecht N, Schmidt S. Measuring mindfulness-the Freiburg Mindfulness Inventory (FMI). Personality and Individual Differences. 2006;40(8):1543-1555. doi:10.1016/j.paid.2005.11.025
- [Background] McConnaughy, E.A., Prochaska, J.O., Velicer, W.F. (1983). Stages of change in psychotherapy: Measurement and sample profiles. Psychotherapy: Theory , Research and Practice, 20 (3) 368-375.
- [Background] University of Rhode Island Change Assessment Scale (URICA): Short Form for Physical Health Behavior State. Accessed June 5, 2022. https://www.camdenhealth.org/wp-content/uploads/2012/10/URICA-Scoring-Guide.docx
- [Background] Condrasky MD, Williams JE, Catalano PM, Griffin SF. Development of psychosocial scales for evaluating the impact of a culinary nutrition education program on cooking and healthful eating. J Nutr Educ Behav. 2011 Nov-Dec;43(6):511-6. doi: 10.1016/j.jneb.2010.09.013. Epub 2011 Aug 15. PMID 21840764
- [Background] RAND Corporation. 36-Item Short Form Survey Instrument (SF-36). Health Care. Accessed June 6, 2022. https://www.rand.org/health-care/surveys_tools/mos/36-item-short-form/survey-instrument.html
- [Background] Wolfson JA, Ishikawa Y, Hosokawa C, Janisch K, Massa J, Eisenberg DM. Gender differences in global estimates of cooking frequency prior to COVID-19. Appetite. 2021 Jun 1;161:105117. doi: 10.1016/j.appet.2021.105117. Epub 2021 Jan 16. PMID 33460693
- [Background] Little RJ, Raghunathan T. On summary measures analysis of the linear mixed effects model for repeated measures when data are not missing completely at random. Stat Med. 1999 Sep 15-30;18(17-18):2465-78. doi: 10.1002/(sici)1097-0258(19990915/30)18:17/183.0.co;2-2. PMID 10474153
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725
- [Background] Wang M, Fitzmaurice GM. A simple imputation method for longitudinal studies with non-ignorable non-responses. Biom J. 2006 Apr;48(2):302-18. doi: 10.1002/bimj.200510188. PMID 16708780
- [Background] Food Research & Action Center. Hunger & Poverty in America. Food Research & Action Center. Accessed June 7, 2022. https://frac.org/hunger-poverty-america
- [Background] Harvard T.H. Chan School of Public Health. "Whole Grains." The Nutrition Source, January 24, 2014. https://www.hsph.harvard.edu/nutritionsource/what-should-you-eat/whole-grains/.